CLINICAL TRIAL: NCT03391882
Title: An Open-Label, Randomized, Crossover Trial Utilizing a Single-Blinded Rater to Evaluate APL-130277 Compared to Subcutaneous Apomorphine in Levodopa Responsive Subjects With Parkinson's Disease Complicated by Motor Fluctuations
Brief Title: A Study of an Investigational Drug to See How it Affects the People With Parkinson's Disease Complicated by Motor Fluctuations ("OFF" Episodes) Compared to an Approved Drug Used to Treat People With Parkinson's Disease Complicated by Motor Fluctuations ("OFF" Episodes)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTH-302; 2016-003456-70 (EudraCT Number)
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Results first posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Motor OFF Episodes Associated With Parkinson's Disease
Keywords: Parkinson's Disease; "Off" Episodes; motor fluctuations associated with Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

STUDY DESIGN:
Masking Description: Open label: APL-130277 and Subcutaneous Apomorphine
  Single-Blinded Rater for MDS-UPDRS Part III Motor Examination assessment in Part B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- APL-130277 (Experimental): APL-130277: Part A- determine the dose; Part B- 28-day repeat dosing at the dose determined in Part A
  Interventions: Drug: APL-130277
- subcutaneous apomorphine (Active Comparator): subcutaneous apomorphine , Part A- determine the dose; Part B- 28-day repeat dosing at the dose determined in Part A
  Interventions: Drug: subcutaneous apomorphine

INTERVENTIONS:
Drug: APL-130277 — APL-130277: Part A- determine the dose; Part B- 28-day repeat dosing at the dose determined in Part A
  Other Names: Apomorphine Hydrochloride
  Arms: APL-130277
Drug: subcutaneous apomorphine — subcutaneous apomorphine Part A- determine the dose; Part B- 28-day repeat dosing at the dose determined in Part A
  Other Names: APO-go®
  Arms: subcutaneous apomorphine

SUMMARY:
A study of an investigational drug to see how it affects the people with Parkinson's Disease complicated by motor fluctuations ("OFF" Episodes) compared to an approved drug used to treat people with Parkinson's Disease complicated by motor fluctuations ("OFF" Episodes)

DETAILED DESCRIPTION:
An Open-Label, Randomized, Crossover Trial utilizing a Single-Blinded Rater to evaluate APL-130277 compared to s.c. Apomorphine in Levodopa Responsive Subjects with Parkinson's Disease Complicated by Motor Fluctuations.

PART A consists of an open label, crossover titration phase where eligible subjects will be randomized to 1 of 2 treatment sequences in a 1:1 ratio to Sublingual APL-130277 followed by subcutaneous apomorphine or subcutaneous apomorphine followed by sublingual APL-130277. Subjects will undergo dose titration with the first study treatment (APL-130277 or sc apomorphine) to tolerance and effect, ie, the tolerable dose that turns the subject from the practically defined "OFF" state to the full "ON" state as determined by both the Investigator and subject. The subject will then be crossed over to the other study treatment (APL-130277 or subcutaneous apomorphine) and similarly titrated to tolerance and effect. These determined doses of APL-130277 and subcutaneous apomorphine will be used during PART B.

PART B consists of an open-label, crossover treatment period where subjects will be randomized to one of the study treatment for 4 weeks, then be crossed over to the other study treatment (APL-130277 or sc apomorphine) for additional 4-weeks of open-label treatment. Subjects return to the clinic for safety and efficacy assessments throughout the treatment period.

This study is designed to test the superiority of sublingually administered APL-130277 against subcutaneously injected apomorphine (APO-go) for the treatment of "OFF" episodes in patients with Parkinson's Disease, as measured by the change from pre-dose to 90 minutes post-dose in MDS UPDRS Part III score in Part B after 4 weeks of dosing in each crossover period.

ELIGIBILITY:
Inclusion Criteria:

1. The subject (and caregiver, if applicable) must be fully informed of and understand the objectives, procedures, and possible benefits and risks of the study, and give written informed consent prior to performing any study related activities.
2. Male or female ≥ 18 years of age.
3. Clinical diagnosis of Idiopathic Parkinson's disease (PD), consistent with UK Brain Bank Criteria (excluding the "more than one affected relative" criterion).
4. Clinically meaningful response to levodopa (L-Dopa), as determined by the Investigator.
5. Subjects at screening must demonstrate an adequate L-Dopa response on the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS UPDRS) Part III in the "ON" state compared to the MDS UPDRS Part III in the "OFF" state and on the Hoehn and Yahr, as determined during the review by Enrollment Adjudication Committee (EAC), Sponsor, and Medical Monitor.
6. Receiving stable doses of L Dopa/carbidopa and/or L Dopa/benserazide and/or L Dopa/carbidopa/entacapone (immediate or chronic release) administered at least 4 times per day OR Rytary™ administered at least 3 times per day for at least 4 weeks before the initial screening Visit (SV1). Adjunctive PD medication regimens are permitted but must be maintained at a stable dose for at least 4 weeks prior to SV1 with the exception of monoamine oxidase B (MAO B) inhibitors, which must be maintained at a stable level for at least 8 weeks prior to SV1.
7. No planned medication change(s) or surgical intervention anticipated during the course of study.
8. Subjects must experience at least one well defined "OFF" episode per day and have a total daily "OFF" time duration of > 2 hours during the waking day, based on judgment of physician and subject self assessment.
9. Subject must have predictable morning "OFF" periods, based on judgment of physician and subject self assessment.
10. Subject, and where appropriate caregiver, must be trained in completing the home dosing diaries and able to recognize "ON" and "OFF" states.
11. Stage III or less on the modified Hoehn and Yahr scale in the "ON" state.
12. Mini-Mental State Examination (MMSE) score > 25.
13. Female subject of childbearing potential and male subject with female partner of childbearing potential must agree to either remain abstinent or use adequate and reliable contraception throughout the study and for at least 7 days after the last dose of study drug has been taken. Note: Continued use of adequate and reliable contraception is recommended through 30 days after study completion.
14. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study related procedures to complete the study.
15. Must be approved as a satisfactory candidate by the Enrollment Adjudication Committee (EAC), Medical Monitor, and Sponsor.

Exclusion Criteria:

1. Atypical or secondary parkinsonism.
2. Major focal brain disorders including malignancy or stroke.
3. Prior treatment with any of the following: a neurosurgical procedure for PD; continuous subcutaneous (subcutaneous) apomorphine infusion; subcutaneous (subcutaneous) apomorphine injection; Duodopa/Duopa; or APL-130277.
4. Contraindications to domperidone, subcutaneous apomorphine, or hypersensitivity to apomorphine hydrochloride or any of the ingredients of subcutaneous apomorphine (notably sodium metabisulfite).
5. Female who is pregnant or lactating.
6. Participation in an interventional clinical study and/or receipt of any investigational (ie, unapproved) medication within 30 days prior to SV1.
7. Currently taking selective 5HT3 antagonists (ie, ondansetron, granisetron, dolasetron, palonosetron, alosetron), dopamine antagonists (excluding quetiapine or clozapine) or dopamine depleting agents. Subjects receiving anti depressants must be on a stable daily dose for at least 8 weeks prior to SV1.
8. The subject has a current diagnosis or history of substance abuse (excluding nicotine and caffeine) or alcohol abuse (in the opinion of the investigator) < 6 months prior to SV1.
9. The recreational use of cannabinoids and hallucinogenic are excluded, as well any use of a sublingual formulation of any drug.
10. Subject has a history of malignancy within 5 years prior to SV1, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
11. Subject has a clinically significant abnormality on screening evaluation including physical examination, vital signs, electrocardiogram (ECG), or laboratory tests that the Investigator considers to be inappropriate to allow participation in the study.
12. Subject has screening laboratory test results of: blood urea nitrogen (BUN) value ≥ 1.5 times the upper limit of normal (ULN) for the reference range; serum creatinine > 1.5 times the ULN for the reference range; or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value ≥ 2 times the ULN for the reference laboratory.
13. Subject has random (non-fasting) screening glucose of ≥ 200 mg/dL (11.1 mmol/L) or HbA1c > 7.0%.
14. Subjects with type 1 diabetes, or insulin dependent diabetics are excluded. Subjects with type 2 diabetes are eligible for study inclusion if the following conditions are met:

    * Subject's screening glucose is < 200 mg/dL (11.1 mmol/L). Note: Subjects with random (non fasting) blood glucose at screening ≥ 200 mg/dL (11.1 mmol/L) must be retested in a fasted state; and
    * Subject's hemoglobin A1c (HbA1c) ≤ 7.0%; and
    * If the subject is currently being treated with oral anti-diabetic medication(s), the dose must have been stable for at least 4 weeks prior to SV1. Such medication may be adjusted or discontinued during the study, as clinically indicated.
15. The subject's screening ECG results of corrected QT interval using Fridericia's formula (QTcF) ≥ 450 msec for male subjects or ≥ 470 msec for female subjects. Eligibility will be based on the core laboratory ECG interpretation report.
16. Subject has a positive screening laboratory test result for human immunodeficiency virus (HIV).
17. Subject has a positive screening laboratory test result for hepatitis B surface antigen or hepatitis C antibodies and has liver function test results at screening above the ULN for the reference laboratory.
18. Subject has any other medical disorder that, in the opinion of the Investigator, could interfere with the subject's participation in the study.
19. Subject has major psychiatric disorder(s), including but not limited to: bipolar disorder, psychosis (eg, Parkinson's Disease Psychosis), major depressive episode, or any disorder that, in the opinion of the Investigator, would require treatment that could make study participation unsafe or make treatment compliance difficult.
20. History of clinically significant impulse control disorder(s).
21. History of symptomatic orthostatic hypotension requiring medication.
22. History of severe dyskinesia based on a score of 4 on the MDS-UPDRS Part IV.
23. Dementia that precludes providing informed consent or would interfere with participation in the study.
24. Current/recent suicidal ideation as evidenced by answering "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at screening (using the "screening /Baseline Version" scale, in the past 12 months) or attempted suicide within the last 5 years.
25. Presence of canker or mouth sores in the 30 days prior to SV1, or other clinically significant oral pathology in the opinion of the Investigator. The Investigator should follow-up with an appropriate specialist on any finding, if indicated, before enrolling a subject into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (31):
- Austria (2):
  - Medical University Innsbruck, Neurolgy Dept, Innsbruck
  - Wilhelminenspital, Department of Neurology, Vienna
- France (2):
  - CHU Caremeau, Service de Neurologie, Nîmes
  - Centre d'Investigation Clinique, CIC 43, CHU Purpan, Hopital Pierre-Paul Riquet, place du Dr. Baylac, Hall D, 2 eme etage -TSA, Toulouse
- Germany (9):
  - Klinken Beelitz GmbH Neurologisches Fachkrankenhaus fur Bewegungsstorungen/Parkinson, Beelitz-Heilstätten
  - Charite-University Medicine Berlin, Department of Neurology, Campus charite Mitte, Berlin
  - St. Joseph Krankenhaus Berlin - Weissensee, Abteilung fur Neurologie, Berlin
  - St. Josef Hospital, Klnikum der Ruhr-Universitat-Bochum, Neurologische Klinik, Bochum
  - Universitatsklinikum Carol Gustav Carus an der TU dDresden, Klinik umd Poliklinik fur Neurologie, Dresden
  - Klinik Haag i.OB, Haag in Oberbayern
  - Curiositas ad sanum GmbH, Munich
  - Klinikum rechts der Isar der Technischen Universitat Munchen, München
  - Universitaets-und Rehabillitatinskliniken Ulm, Ulm
- Italy (6):
  - San Raffaele Cassino, Cassino
  - University Hospital Policlinico-Vittorio Emanuele, Department "G.F. Ingrassia", Section of Neurosciences, Catania
  - A.O.U. Universita degli Studi della Campania "Luigi Vanvitelli" Dipartamento di Scienze Mediche e Chirurgiche Avanzate, Napoli
  - IRCCS San Raffaele Pisana-Clinical Trial Center, Rome
  - Istituto Clinico Humanitas, Dipartmento di Neurologia 1, Rozzano
  - AOU San Giovanni di Dio e Ruggid'Aragona-CEMAND, Salerno
- Spain (7):
  - Hospital Universitario de Cruces, Neurology, Barakaldo
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau c/Mas de Casanovas 90, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario de la Princesa, Madrid
  - CINAC, Hospital Universitario HB Pueta del Sur, Móstoles
  - Hospital General de Catalunya, Sant Cugat del Vallès
- United Kingdom (5):
  - King's College Hospital NHS Foundation Trust, London
  - 10W, Imperial Memory/PD Research Unit, Imperial College Healthcare NHS Trust, London
  - NHS Forth Valley, Pennine Actue NHS Trust, Fairfield General Hospital, Manchester
  - Academic Neuroscience Department, C Floor, South Block, Nottingham University Hospitals NHS Trust Queens Medical Centre, Nottingham
  - University Hospitals Plymouth NHS Trust-Derriford Hospital-The Lind Research Center, Level 5, Terence Lewis Building, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Individual Patient Data (IPD) for this study may be made available upon request via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be made available upon request within 12 months of posting the study results on ct.gov.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- APL-SC: Part A - Titration Phase: APL (APL-130277) then SC (subcutaneous apomorphine); Did not continue in Part B - Treatment Phase.
- SC-APL: Part A - Titration Phase: SC (subcutaneous apomorphine) then apomorphine hydrochloride APL (APL-130277); Did not continue in Part B - Treatment Phase.
- APL-SC-APL-SC: Part A - Titration Phase: APL (APL-130277) then SC (subcutaneous apomorphine) into Part B - Treatment Phase: APL then SC
- APL-SC-SC-APL: Part A - Titration Phase: APL (APL-130277) then SC (subcutaneous apomorphine); Randomized into Part B - Treatment Phase: SC then APL
- SC-APL-APL-SC: Part A - Titration Phase: SC (subcutaneous apomorphine) then APL (APL-130277); Randomized into Part B - Treatment Phase: APL then SC
- SC-APL-SC-APL: Part A - Titration Phase: SC (subcutaneous apomorphine) then APL (APL-130277); Randomized into Part B - Treatment Phase: SC then APL
Period: Study Overall
Arm/Group | APL-SC | SC-APL | APL-SC-APL-SC | APL-SC-SC-APL | SC-APL-APL-SC | SC-APL-SC-APL
Started | 20 | 19 | 19 | 18 | 18 | 19
Safety Population | 20 | 18 | 19 | 18 | 18 | 19
Modified Intent-to-Treat Population | 20 | 18 | 19 | 18 | 18 | 19
Completed (The study) | 0 | 0 | 16 | 15 | 14 | 15
Not Completed | 20 | 19 | 3 | 3 | 4 | 4
Not completed — Adverse Event | 3 | 6 | 1 | 1 | 3 | 1
Not completed — Lack of Efficacy | 13 | 9 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 2 | 2 | 1 | 3
Not completed — EARLY TERM AT SPONSOR REQUEST | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Period: Part A - Titration Phase
Arm/Group | APL-SC | SC-APL | APL-SC-APL-SC | APL-SC-SC-APL | SC-APL-APL-SC | SC-APL-SC-APL
Started | 20 | 19 | 19 | 18 | 18 | 19
Safety Population Part A | 20 | 18 | 19 | 18 | 18 | 19
Modified Intent-to-Treat Population Part A | 20 | 18 | 19 | 18 | 18 | 19
Completed (Part A) | 2 | 3 | 19 | 18 | 18 | 19
Not Completed | 18 | 16 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 6 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 12 | 6 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0 | 0 | 0 | 0
Not completed — EARLY TERM AT SPONSOR REQUEST | 0 | 1 | 0 | 0 | 0 | 0
Period: Post Part A / Pre Part B
Arm/Group | APL-SC | SC-APL | APL-SC-APL-SC | APL-SC-SC-APL | SC-APL-APL-SC | SC-APL-SC-APL
Started | 2 | 3 | 19 | 18 | 18 | 19
Completed | 0 | 0 | 19 | 18 | 18 | 19
Not Completed | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Period: Part B - Treatment Phase
Arm/Group | APL-SC | SC-APL | APL-SC-APL-SC | APL-SC-SC-APL | SC-APL-APL-SC | SC-APL-SC-APL
Started | 0 | 0 | 19 | 18 | 18 | 19
Safety Population Part B | 0 | 0 | 19 | 18 | 18 | 19
Modified Intent-to-Treat Population Part B | 0 | 0 | 19 | 18 | 18 | 19
Completed (Part B) | 0 | 0 | 16 | 15 | 14 | 15
Not Completed | 0 | 0 | 3 | 3 | 4 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | APL-SC | SC-APL | APL-SC-APL-SC | APL-SC-SC-APL | SC-APL-APL-SC | SC-APL-SC-APL | Total
Number analyzed (Participants) | 20 | 18 | 19 | 18 | 18 | 19 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 8 | 10 | 9 | 8 | 52
  >=65 years | 11 | 10 | 11 | 8 | 9 | 11 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (8.33) | 63.9 (9.99) | 65.0 (9.80) | 63.2 (6.91) | 63.4 (9.71) | 65.6 (8.69) | 64.4 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 6 | 1 | 6 | 7 | 34
  Male | 13 | 11 | 13 | 17 | 12 | 12 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 1 | 1 | 2 | 1 | 8
  Not Hispanic or Latino | 19 | 15 | 18 | 16 | 16 | 18 | 102
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 20 | 18 | 19 | 18 | 18 | 19 | 112
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Country [Count of Participants; unit: Participants]
  Austria | 1 | 0 | 2 | 1 | 1 | 0 | 5
  Germany | 6 | 2 | 8 | 10 | 5 | 10 | 41
  Spain | 7 | 8 | 4 | 3 | 5 | 4 | 31
  France | 1 | 1 | 0 | 0 | 0 | 1 | 3
  United Kingdom | 1 | 1 | 1 | 3 | 2 | 3 | 11
  Italy | 4 | 6 | 4 | 1 | 5 | 1 | 21
Baseline Height (cm) [Mean (Standard Deviation); unit: cm] | 168.05 (12.626) | 165.62 (12.348) | 171.91 (10.260) | 174.78 (6.632) | 170.94 (9.795) | 171.16 (9.929) | 170.39 (10.652)
Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] | 74.25 (16.151) | 70.91 (18.624) | 78.45 (21.893) | 80.31 (11.691) | 83.26 (24.383) | 77.14 (15.284) | 77.34 (18.470)
Baseline BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.19 (4.436) | 25.60 (4.813) | 26.36 (5.866) | 26.34 (4.013) | 28.12 (6.100) | 26.30 (4.912) | 26.48 (5.016)
Apomorphine naive at screening [Count of Participants; unit: Participants]
  N | 1 | 2 | 5 | 2 | 2 | 1 | 13
  Y | 19 | 16 | 14 | 16 | 16 | 18 | 99
Total Daily Levodopa Dose Category (mg) [Count of Participants; unit: Participants]
  < 900 mg | 15 | 13 | 15 | 14 | 15 | 14 | 86
  >= 900 mg | 5 | 5 | 4 | 4 | 3 | 5 | 26
Parkinson's disease duration Group [Count of Participants; unit: Participants]
  <=10 years | 17 | 14 | 11 | 12 | 10 | 11 | 75
  >10 years | 3 | 4 | 8 | 6 | 8 | 8 | 37
Movement Disorders Society Unified Parkinson Part III Score assessed prior to levodopa dosing at SV2 [Mean (Standard Deviation); unit: Units on a scale] — The summary score used here is Part III motor examination score. Each Part III item has a 0-4 rating, where 0=normal, 1=slight, 2=mild, 3= moderate, and 4=severe. Higher MDS-UPDRS scores reflect worse motor function. MDS-UPDRS III is a total of 18 questions with 33 individual items, each item ranges from 0-4. The MDS-UPDRS III motor score is the summation of all these 33 individual item scores, and hence ranges from 0-132. Score drops over time imply improvement in motor function (higher values represent a worse outcome). SV2= Screening Visit 2
  Units on a scale | 53.6 (13.11) | 50.6 (14.74) | 50.3 (12.18) | 50.1 (10.33) | 53.3 (15.20) | 48.6 (13.36) | 51.1 (13.07)
Change in MDS-UPDRS Part III Score from Pre-dose to 30 minutes after levodopa dosing at SV2 [Mean (Standard Deviation); unit: Units on a scale] — The summary score used here is Part III motor examination score. Each Part III item has a 0-4 rating, where 0=normal, 1=slight, 2=mild, 3= moderate, and 4=severe. Higher MDS-UPDRS scores reflect worse motor function. MDS-UPDRS III is a total of 18 questions with 33 individual items, each item ranges from 0-4. The MDS-UPDRS III motor score is the summation of all these 33 individual item scores, and hence ranges from 0-132. Score drops over time imply improvement in motor function (higher values represent a worse outcome). SV2= Screening Visit 2 Population: safety population
  Units on a scale
    number analyzed (Participants) | 19 | 18 | 19 | 18 | 17 | 19 | 110
    (all) | -18.0 (12.33) | -16.2 (11.80) | -19.8 (13.64) | -22.9 (12.09) | -21.9 (14.19) | -21.8 (12.53) | -20.1 (12.70)

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-dose to 90 Mins. Post-dose in Movement Disorders Society Unified Parkinson's Disease Rating Scale Part III Score After 4 Weeks of Dosing in Each Crossover Period (Assessed by the Blinded-rater In-clinic at Visit 3 and Visit 6 of PART B).
Description: The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a clinimetric assessment of subjective and objective symptoms and signs of Parkinson's disease created by the Movement Disorder Society. The summary score used in this study for the primary objective and primary efficacy endpoint is Part III motor examination score. Each Part III item has a 0-4 rating, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. Higher MDS-UPDRS scores reflect worse motor function. MDS-UPDRS III is a total of 18 questions with 33 individual items, each item ranges from 0-4. The MDS-UPDRS III motor score is the summation of all these 33 individual item scores, and hence ranges from 0-132. Score drops over time imply improvement in motor function (higher values represent a worse outcome).
Time Frame: Pre-dose to 90 minutes post-dose at Week 4 of each treatment period (Visit 3 and 6)
Population: Part B mITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- SC (Subcutaneous Apomorphine): subcutaneous apomorphine
- APL (APL-130277): APL-130277
Arm/Group | SC (Subcutaneous Apomorphine) | APL (APL-130277)
Number analyzed (Participants) | 61 | 62
Units on a scale | -13.78 [-16.65 to -10.90] | -13.55 [-16.39 to -10.70]
Statistical Analysis 1: Comparison: SC (Subcutaneous Apomorphine) vs APL (APL-130277); Test type: Superiority; p = 0.8944, Mixed Models Analysis; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-3.16 to 3.62], Standard Error of Mean 1.722

2. Secondary Outcome: Durability of Effect, Defined as an Investigator Confirmed Full "ON" Within 30 Minutes Post Dose and at 90 Minutes Post-dose, After 4 Weeks of Dosing in Each Crossover Period (Assessed by the Blinded-rater In-clinic at Visit 3 and Visit 6 of PART B).
Description: Investigator will confirm whether subject is "OFF", Full "ON" or Partial "ON" , and note the time the subject changes from "OFF" to Partial "ON" or Full "ON". The Investigator will also record the subject "ON"/"OFF" status (binary variable, Yes / No) prior to performing each MDS-UPDRS Part III assessment. Durability of effect is defined as an Investigator confirmed full "ON" within 30 minutes post-dose and at 90 minutes post-dose, after 4 weeks of dosing in each PART B crossover period.
  Response rate = % of subjects that achived full "ON" within the timeframe
Time Frame: Within 30 minutes post-dose and at 90 minutes post-dose at Week 4 of each treatment period (Visit 3 and 6)
Population: Part B mITT population
Measure: Number; unit: Percentage of participants
Groups:
- APL (APL-130227): APL-130227
Arm/Group | SC (Subcutaneous Apomorphine) | APL (APL-130227)
Number analyzed (Participants) | 61 | 62
Percentage of participants | 18.03 | 17.74
Statistical Analysis 1: Comparison: SC (Subcutaneous Apomorphine) vs APL (APL-130227); Test type: Superiority; p = 0.7777, generalized linear random effects model; Odds Ratio (OR) = 1.129, 95% CI 2-sided [0.484 to 2.637]

3. Secondary Outcome: Subject Preference for APL Treatment as Measured by the Subject Treatment Preference Questionnaire (TPQ), Planned After the Subject Had Completed Both APL-130277 and sc Apomorphine Treatment Regimens (Assessed In-clinic at Visit 6 of PART B)
Description: The TPQ assessment of subject treatment preference was changed from being based on a visual analogue scale or VAS (Q9b)) to a 5-point Likert scale (Q9a). Subject reported preference for APL or SC was based on question Q9a or Q9b combined. For Q9a, responses were dichotomized as follows for statistical analysis: preference for APL (responses of either definitely or somewhat prefer APL) versus no preference for APL (responses of no preference, or somewhat/definitely prefer sc apomorphine). The VAS score was similarly dichotomized as preference for APL (score of >0 to 50) versus no preference for APL (-50 to 0). If a subject responded to both Q9a and Q9b, then Q9a only was used.
Time Frame: After 8 weeks of treatment (Visit 6)
Population: Part B mITT population
Measure: Number (95% Confidence Interval); unit: % of participants
Groups:
- Overall: Overall
Arm/Group | Overall
Number analyzed (Participants) | 72
% of participants | 72.2 [61.9 to 82.6]
Statistical Analysis 1: Comparison: Overall; Test type: Superiority; p = 0.0002, binomial distribution with normal approx — The p-value is from a 1-sample, 2-sided test of the null hypothesis that the true proportion preferring APL is 50% to evaluate if a significantly higher proportion of the subjects prefer APL-130277 or not

4. Secondary Outcome: Subject Confirmed Durability of Effect, Defined as Subject Confirmed Full "ON" Within 30 Minutes Post-dose and at 90 Minutes Post-dose, After 4 Weeks of Dosing in Each Crossover Period (Assessed In-clinic at Visit 3 and Visit 6 of PART B).
Description: Patients will confirm whether he/she is "OFF", Full "ON" or Partial "ON", and the staff will ask the subject to notify the staff when he/she changes from "OFF" to Partial "ON" or Full "ON" (binary variable, Yes / No) . Subject confirmed durability of effect is defined as subject confirmed full "ON" within 30 minutes post-dose and at 90 minutes post-dose, after 4 weeks of dosing in each crossover period (assessed in-clinic at V3 and V6 of PART B).
  Response rate = % subjects that achived full ON within the timeframe
Time Frame: Week 4
Population: Part B mITT population
Measure: Number; unit: Percentage of participants
Arm/Group | SC (Subcutaneous Apomorphine) | APL (APL-130227)
Number analyzed (Participants) | 61 | 62
Percentage of participants | 14.75 | 19.36
Statistical Analysis 1: Comparison: SC (Subcutaneous Apomorphine) vs APL (APL-130227); Test type: Superiority; p = 0.1769, generalized linear random effects model; Odds Ratio (OR) = 1.835, 95% CI 2-sided [0.759 to 4.438]

5. Secondary Outcome: Patient Global Impression of Change (PGI-C): Subject Improvement of "OFF" Episodes, Defined as Very Much Better, Much Better or a Little Better After 4 Weeks of Dosing in Each Crossover Period (Assessed In-clinic at Visit 3 and Visit 6 of PART B).
Description: The PGI-C is the patient reported outcome counterpart to the Clinical Global Impressions scale, (CGI), which was published in 1976 by the National Institute of Mental Health (US). It consists of one item taken from the CGI and adapted to the patient. The PGI-C is based on a 7-point scale, where a lower score is associated with higher symptom improvement. The scale is:
  Very much better Much better A little better No change A little worse Much worse Very much worse
  Subject improvement of "OFF" episodes is defined as very much better, much better or a little better at Week 4 in each PART B crossover period.
  Response rate= % of subjects who achieved improvement of "OFF" episodes
Time Frame: At Week 4 of each treatment period (Visit 3 and 6, or Early Termination)
Population: Part B mITT population
Measure: Number; unit: Percentage of participants
Arm/Group | SC (Subcutaneous Apomorphine) | APL (APL-130277)
Number analyzed (Participants) | 70 | 71
Percentage of participants | 77.14 | 83.10
Statistical Analysis 1: Comparison: SC (Subcutaneous Apomorphine) vs APL (APL-130277); Test type: Superiority; p = 0.3922, generalized linear random effects model; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.61 to 3.53]

ADVERSE EVENTS:
Time Frame: 10 weeks (from first dose of study drug to last study visit)
Groups:
- Part A Dose Titration: APL (APL-130277): Part A Dose Titration: APL (APL-130277)
- Part A Dose Titration: SC (Subcutaneous Apomorphine): Part A Dose Titration: SC (Subcutaneous Apomorphine)
- Part B Treatment: APL (APL-130277): Part B Treatment: APL (APL-130277)
- Part B Treatment: SC (Subcutaneous Apomorphine): Part B Treatment: SC (Subcutaneous Apomorphine)
Arm/Group | Part A Dose Titration: APL (APL-130277) | Part A Dose Titration: SC (Subcutaneous Apomorphine) | Part B Treatment: APL (APL-130277) | Part B Treatment: SC (Subcutaneous Apomorphine)
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/97 | 0/71 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/102 | 1/97 | 1/71 | 1/70
Other Adverse Events (participants affected / at risk) | 52/102 | 44/97 | 23/71 | 37/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Dose Titration: APL (APL-130277) (N=102) | Part A Dose Titration: SC (Subcutaneous Apomorphine) (N=97) | Part B Treatment: APL (APL-130277) (N=71) | Part B Treatment: SC (Subcutaneous Apomorphine) (N=70)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Dose Titration: APL (APL-130277) (N=102) | Part A Dose Titration: SC (Subcutaneous Apomorphine) (N=97) | Part B Treatment: APL (APL-130277) (N=71) | Part B Treatment: SC (Subcutaneous Apomorphine) (N=70)
Nausea (Gastrointestinal disorders) | 32 (53) | 22 (31) | 10 (25) | 11 (21)
Fatigue (General disorders) | 6 (6) | 10 (10) | 4 (4) | 4 (5)
Injection site erythema (General disorders) | 0 (0) | 6 (9) | 1 (1) | 5 (5)
Injection site haematoma (General disorders) | 0 (0) | 2 (2) | 0 (0) | 19 (23)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 4 (5) | 1 (3)
Dizziness (Nervous system disorders) | 10 (15) | 4 (4) | 2 (2) | 3 (3)
Dyskinesia (Nervous system disorders) | 8 (10) | 7 (13) | 8 (11) | 14 (20)
Somnolence (Nervous system disorders) | 9 (9) | 13 (18) | 3 (3) | 4 (4)
Yawning (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (8) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 4 (5) | 5 (5) | 3 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03391882/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03391882/SAP_001.pdf